CLINICAL TRIAL: NCT00508300
Title: Epidural Analgesia (EDA) Versus Patient Controlled Analgesia (PCA) in Laparoscopic Colon Surgery: A Monocentric Controlled Non-blinded Randomized Superiority Trial
Brief Title: Epidural Analgesia (EDA) Versus Patient Controlled Analgesia (PCA) in Laparoscopic Colon Surgery
Acronym: EVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, professor of surgery, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P166/07
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Laparoscopic Colectomy
Keywords: laparoscopic; colectomy; Fast Track; epidural
MeSH Terms: interventions — Analgesia, Epidural; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Epidural Analgesia (EDA) An epidural catheter was inserted at thoracic level (Th8-Th10) before induction of anesthesia. A bolus of 5 mL of bupivacaine 0.5% was started as soon as the epidural catheter was in place, and a continuous perfusion of bupivacaine 0.5% at 5 mL/hr was initiated until the end of surgical procedure.
  Interventions: Procedure: Epidural analgesia
- B (Other): Patient controlled analgesia (PCA) was assured by fentanyl (morphine-based) as needed.
  Interventions: Procedure: Patient controlled analgesia

INTERVENTIONS:
Procedure: Epidural analgesia — Thoracic epidural analgesia until day 2
  Arms: A
Procedure: Patient controlled analgesia — Patient controlled analgesia (morphine-based)
  Arms: B

SUMMARY:
The purpose of this study is to determine whether a epidural analgesia versus patient controlled analgesia reduces the medical recovery in patients undergoing elective laparoscopic colon surgery.

DETAILED DESCRIPTION:
Allocation by individual random number generated by a computer program to either EDA or PCA for 48h after laparoscopic colonic surgery.

Short, both groups are treated according to a recent Fast track protocol. Group A will preoperatively receive a mid thoracic EDA (th 8-9; naropine 0,1%) while group B will receive a PCA (morphine) postoperatively. Both EDA and PCA are removed the afternoon at day 2. Patients with a non-functioning EDA within the first 24h will be crossed over to the PCA group.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for elective laparoscopic colonic surgery

Exclusion Criteria:

* Age < 18y
* No informed consent
* Emergency situation
* Contraindication for EDA (according to local Anesthesia guidelines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Demartines, MD, Study Chair — Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland
Locations (1):
- Department of Visceral Surgery, University Hospital CHUV, Lausanne, Lausanne, Switzerland

REFERENCES:
- [Derived] Hubner M, Blanc C, Roulin D, Winiker M, Gander S, Demartines N. Randomized clinical trial on epidural versus patient-controlled analgesia for laparoscopic colorectal surgery within an enhanced recovery pathway. Ann Surg. 2015 Apr;261(4):648-53. doi: 10.1097/SLA.0000000000000838. PMID 25119117

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural: Epidural Analgesia (Th 8-9)
  Epidural analgesia: Thoracic epidural analgesia until day 2
- Patient-controlled Analgesia: Patient controlled analgesia (morphine-based)
  Patient controlled analgesia: Patient controlled analgesia (morphine-based)
Period: Overall Study
Arm/Group | Epidural | Patient-controlled Analgesia
Started | 67 | 61
Completed | 65 | 57
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: 128 patients were randomized to receive either EDA (n = 67) or PCA (n = 61) as allocated treatment. Two EDA patients and our PCA patients dropped out after randomization and no patient was lost to follow-up. Final analysis compared therefore 65 EDA patients with 57 PCA patients (Fig. 1).
Groups:
- Epidural: epidural catheter was inserted at thoracic level (Th8-Th10) before induction of anesthesia. A bolus of 5 mL of bupivacaine 0.5% was started as soon as the epidural catheter was in place, and a continuous perfusion of bupivacaine 0.5% at 5 mL/hr was initiated until the end of surgical procedure.
- Patient-controlled Analgesia: In the PCA group, intravenous PCA was inserted with 1 mg/h. A bolus of 1 mL was allowed at every 5 minutes up to a maximal dose of 40 mg/4h.
- Total: Total of all reporting groups
Arm/Group | Epidural | Patient-controlled Analgesia | Total
Number analyzed (Participants) | 65 | 57 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (15.1) | 61.2 (17.8) | 62.5 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 37 | 34 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 65 | 57 | 122

OUTCOME MEASURES:

1. Primary Outcome: Medical Recovery (Defined as Pain Sufficient Controlled by Oral Analgesia, Fully Mobile Patients or at Least as Mobile as at Admission and Tolerance of the Patient of Oral Food Intake (More Than 2/3 of Daily Meal))
Description: Medical recovery was chosen as primary end point and was defined as the fulfillment of all the 3 following criteria: (1) sufficient pain control by oral analgesics, (2) fully mobilized or at least comparable with preoperative status, and (3) tolerance of oral food that was defined as two thirds or more of normal meal (hospital portion).23 Medical recovery was considered as more specific outcome parameter than hospital stay because social and logistic factors were not interfering.24,25
Time Frame: 30 days
Population: accorindg to intention-to-treat principle
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Epidural | Patient-controlled Analgesia
Number analyzed (Participants) | 65 | 57
days | 5 [3 to 7.5] | 4 [3 to 6]

2. Secondary Outcome: Complication Rate, Peridural Analgesia Failure Rate, Patient Comfort
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until 30 days after surgery.
Arm/Group | Epidural | Patient-controlled Analgesia
All-Cause Mortality (participants affected / at risk) | 2/65 | 0/57
Serious Adverse Events (participants affected / at risk) | 13/65 | 5/57
Other Adverse Events (participants affected / at risk) | 0/65 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural (N=65) | Patient-controlled Analgesia (N=57)
major complications according to clavien: 3+4 (Surgical and medical procedures) | 13 (13) | 5 (5) — clavien 3+4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes